CLINICAL TRIAL: NCT07198165
Title: Short-Course Radiotherapy Combined With CAPOX and Bevacizumab, With or Without PD-1 Inhibitors, as Total Neoadjuvant Therapy for Locally Advanced Rectal Cancer
Brief Title: SCRT Followed by CAPOX + Bev ± PD-1 Inhibitor for TNT in LARC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Bo Feng, Chief Physician, Ruijin Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TRAINER-2
Record Dates: First submitted 2025-09-21; First posted 2025-09-30 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Rectal Cancer; Rectal Adenocarcinoma; Rectal Cancer, Radiotherapy; Rectal Cancer Patients; Immunotherapy; Total Neoadjuvant Therapy; Total Neoadjuvant Treatment; Targeted Therapy; Chemoradiotherapy
Keywords: Rectal cancer; Total Neoadjuvant Therapy; Immunotherapy; Targeted therapy; Chemoradiotherapy
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (No Intervention): Short-course radiotherapy (25Gy/5Fx) followed by 4 cycles of CAPOX regimen (Oxaliplatin 130mg/m² IV infusion, Capecitabine 1000mg/m² orally for 14 days, Q3w) combined with Bevacizumab (7.5mg/kg IV infusion, D1, Q3w) .Following completion of total neoadjuvant therapy, the treatment strategy (watch-and-wait or surgical resection) will be selected based on tumor response. The decision regarding adjuvant chemotherapy will be determined according to postoperative pathological findings.
- Intervention group (Experimental): Short-course radiotherapy (25Gy/5Fx) followed by 4 cycles of CAPOX regimen (Oxaliplatin 130mg/m² IV infusion, Capecitabine 1000mg/m² orally for 14 days, Q3w) combined with Bevacizumab (7.5mg/kg IV infusion, D1, Q3w) + PD-1 inhibitor (Toripalimab 240mg IV infusion, D1, Q3w). Following completion of total neoadjuvant therapy, the treatment strategy (watch-and-wait or surgical resection) will be selected based on tumor response. The decision regarding adjuvant chemotherapy will be determined according to postoperative pathological findings.
  Interventions: Drug: PD-1 inhibitor based immunotherapy

INTERVENTIONS:
Drug: PD-1 inhibitor based immunotherapy — Short-course radiotherapy (25Gy/5Fx) followed by 4 cycles of CAPOX regimen (Oxaliplatin 130mg/m² IV infusion, Capecitabine 1000mg/m² orally for 14 days, Q3w) combined with Bevacizumab (7.5mg/kg IV infusion, D1, Q3w) + PD-1 inhibitor (Toripalimab 240mg IV infusion, D1, Q3w).
  Arms: Intervention group

SUMMARY:
This study aims to evaluate the efficacy and safety of short-course radiotherapy combined with CAPOX plus bevacizumab with or without a PD-1 inhibitor in patients with locally advanced rectal cancer (LARC). The hypothesis is that the addition of immunotherapy (PD-1 inhibitor) can significantly improve the complete response (CR) rate and enhance local control while reducing the incidence of distant metastasis. This study will compare the effects of sequential chemoradiotherapy and targeted therapy with or without immunotherapy following short-course radiotherapy, aiming to explore the optimal regimen for total neoadjuvant therapy.

ELIGIBILITY:
Inclusion Criteria:

* Histopathologically confirmed rectal adenocarcinoma with no prior antitumor therapy.
* Exclusion of patients with BRAF mutations or MSI-H status, as determined by pre-enrollment genetic testing including RAS, BRAF, and MSI analysis. RAS mutation status is permitted regardless.
* Absence of severe intestinal obstruction symptoms and no evidence of distant metastasis confirmed by imaging examinations such as CT, MRI, or PET/CT.
* Confirmation as locally advanced rectal cancer by rectal MRI, meeting one or more of the following criteria: T3c-d or T4, N2, EMVI(+), MRF(+), lateral lymph node metastasis; or patients with low-lying rectal cancer (≤5 cm from the anal verge) unsuitable for sphincter-preserving surgery prior to neoadjuvant therapy.
* Age 18 to 75 years.
* ECOG Performance Status of 0 to 1, without severe comorbid medical conditions.
* Adequate organ function:

Hematopoietic: Hemoglobin ≥90 g/L, Platelets ≥80 × 10^9/L, Absolute Neutrophil Count ≥1.5 × 10^9/L.

Hepatic: ALT and AST < 2.5 × ULN. Renal: Serum Creatinine < 1.5 × ULN.

* Provision of signed and dated written informed consent.

Exclusion Criteria:

* Patients found to have BRAF mutations or MSI-H status.
* Patients who have previously received chemotherapy, radiotherapy, immunotherapy, targeted therapy, or surgical resection for colorectal cancer prior to enrollment.
* History or presence of another malignancy (except for early-stage basal cell carcinoma or carcinoma in situ of the cervix) within the past 3 years, with the disease not under control.
* Patients who are pregnant (confirmed by serum or urine β-HCG test) or breastfeeding.
* Patients with severe cardiac, hepatic, renal, neurological, or psychiatric diseases.
* Patients with active infections.
* Poor overall health status, with an ECOG performance status ≥2.
* Patients who have undergone organ transplantation requiring immunosuppressive therapy, or those requiring long-term corticosteroid treatment for autoimmune diseases.
* Patients with comorbid conditions that, in the investigator's judgment, seriously endanger the patient's safety or affect the completion of the study.
* Known hypersensitivity to any of the study drugs.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2025-09-05 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Complete Response rate | 2 weeks after the surgery
  Measurement Methods:
  Chi-square test, Fisher's exact test, multivariate regression analysis (Cox regression model).
  Description:
  For pCR and cCR, chi-square test or Fisher's exact test was used to compare differences between the two groups. Multivariate regression analysis (Cox regression model) was employed to assess the relationship between the intervention and the CR rate.

SECONDARY OUTCOMES:
Disease-Free Survival (DFS) | from enrollment to the end of follow-up at 48 months
  Measurement Method:
  Kaplan-Meier survival analysis, Log-rank test to compare survival curves between the two groups.
  Methods for Handling Missing Values:
  * For missing data, the Last Observation Carried Forward (LOCF) method or multiple imputation method will be applied.
  * For subjects with significant non-compliance or loss to follow-up, sensitivity analysis will be considered to assess the impact on results.
Distant Metastasis Rate | from enrollment to the end of follow-up at 48 months
  Measurement Method:
  Kaplan-Meier survival analysis, Log-rank test to compare survival curves between the two groups.
  Methods for Handling Missing Values:
  * For missing data, the Last Observation Carried Forward (LOCF) method or multiple imputation method will be applied.
  * For subjects with significant non-compliance or loss to follow-up, sensitivity analysis will be considered to assess the impact on results.
Local Recurrence Rate | from enrollment to the end of follow-up at 48 months
  Measurement Method:
  Kaplan-Meier survival analysis, Log-rank test to compare survival curves between the two groups.
  Methods for Handling Missing Values:
  * For missing data, the Last Observation Carried Forward (LOCF) method or multiple imputation method will be applied.
  * For subjects with significant non-compliance or loss to follow-up, sensitivity analysis will be considered to assess the impact on results.
Overall Survival (OS) | from enrollment to the end of follow-up at 48 months
  Measurement Method:
  Kaplan-Meier survival analysis, Log-rank test to compare survival curves between the two groups.
  Methods for Handling Missing Values:
  * For missing data, the Last Observation Carried Forward (LOCF) method or multiple imputation method will be applied.
  * For subjects with significant non-compliance or loss to follow-up, sensitivity analysis will be considered to assess the impact on results.
Pathological Stage | 2 weeks after the surgery
  ypT and ypN staging
  Measurement Method:
  Chi-square test or Fisher's exact test
Tumor Regression Grade(TRG) | 2 weeks after the surgery
  Measurement Method:
  Chi-square test or Fisher's exact test
Sphincter Preservation Rate | 2 weeks after the surgery
  Measurement Method:
  Logistic regression analysis
  Methods for Handling Missing Values:
  * For missing data, the Last Observation Carried Forward (LOCF) method or multiple imputation method will be applied.
  * For subjects with significant non-compliance or loss to follow-up, sensitivity analysis will be considered to assess the impact on results.

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, China

IPD SHARING:
Plan to Share IPD: No